CLINICAL TRIAL: NCT00479492
Title: A 12-Week, Randomized, Subject And Investigator Blind, Placebo-Controlled Trial To Evaluate The Effect Of CP-866,087 On Weight Loss In Obese, Otherwise Healthy Adult Subjects
Brief Title: Study To Determine The Effects And Safety Of A Weight Loss Compound On Overweight, Otherwise Healthy, Volunteers
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Director, Clinical Trial Disclosure Group, Pfizer, Inc.
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: A5051019
Record Dates: First submitted 2007-05-24; First posted 2007-05-28 (Estimated); Last update posted 2009-10-01 (Estimated); Status verified 2008-10

CONDITIONS: Obesity
Keywords: Obesity, weight loss
MeSH Terms: conditions — Obesity; Weight Loss | interventions — CP-866,087

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- 1 (Experimental)
  Interventions: Drug: CP-866,087
- 2 (Experimental)
  Interventions: Drug: CP-866,087
- 3 (Experimental)
  Interventions: Drug: CP-866,087
- 4 (Placebo Comparator)
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: CP-866,087 — 1 mg of CP-866,087, administered QD for 84 days
  Arms: 1
Drug: CP-866,087 — 5 mg of CP-866,087, administered QD for 84 days
  Arms: 2
Drug: CP-866,087 — 10 mg of CP-866,087, administered QD for 84 days
  Arms: 3
Drug: placebo — placebo administered QD for 84 days
  Arms: 4

SUMMARY:
The purpose of this study is to determine whether CP-866,087 is effective in the weight loss of overweight patients.

ELIGIBILITY:
Inclusion Criteria:

* Body Mass Index (BMI) 30 to 40 kg/m2 and total body weight of >110 lbs.
* Otherwise healthy

Exclusion Criteria:

* Women must be of non-childbearing potential.
* Significant current or history of medical illness.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 94 (Actual)
Dates: Start 2007-06; Primary Completion 2008-01 (Actual); Study Completion 2008-01 (Actual)

PRIMARY OUTCOMES:
Measure the effect of weight loss over 12 weeks in overweight otherwise healthy patients. Measurements will include body weight and waist circumference. Measurements will occur at Day 1, 7, 14, 28, 42, 56, 70, 84 and 94. | 94 days

SECONDARY OUTCOMES:
To characterize the effect of 4 weeks of dosing of 3 different doses of CP-866,087 on 24-hour urinary cortisol levels. Measured at Day 1 and Day 29 | 29 days
Exploratory biomarkers measured at Day 1, 14, 28, 56, and 84. | 84 days
Waist circumference measured at Day 1, 7, 14, 28, 42, 56, 70, 84, 94. | 94 days
To explore changes in pharmacodynamics (PD) markers of efficacy resulting from multiple PO doses of CP-866,087, including waist circumference, and serum lipids and exploratory biomarkers. | 94 days
Serum Lipids measured at Day 1, 7, 14, 28, 56, 84 and 94. | 94 days
To explore the effects of chronic, 12-week dosing with CP-866,087 on neuroendocrine endpoints, including testosterone, TSH, T4, and IGF1. Measured at Day 1, 28, 84 and 94. | 94 days

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (4):
- United States (4):
  - Pfizer Investigational Site, Orlando, Florida
  - Pfizer Investigational Site, Kalamazoo, Michigan
  - Pfizer Investigational Site, Portland, Oregon
  - Pfizer Investigational Site, San Antonio, Texas

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A5051019&StudyName=Study%20To%20Determine%20The%20Effects%20And%20Safety%20Of%20A%20Weight%20Loss%20Compound%20On%20Overweight%2C%20Otherwise%20Healthy%2C%20Volunteers